CLINICAL TRIAL: NCT04764630
Title: Clinical Study to Investigate the Pharmacokinetics of Multiple Repeated Doses of Intranasal Naloxone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SCR-011
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Healthy Subjects; Opioid Antagonist; Pharmacokinetics
Keywords: Opioid antagonist; Intranasal naloxone; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This is a three-way crossover study where subjects will be randomized to one of six possible treatment sequences.
Masking Description: The study will be unblinded as the product is administered intranasally and different arms will have a different number of administrations at different times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- A. Four naloxone nasal spray doses (1 every 2.5 min) (Experimental): Four 4 mg IN naloxone doses (left nostril at 0 min, right nostril at 2.5 min, left nostril at 5 min, right nostril at 7.5 min)
  Interventions: Drug: Four naloxone nasal spray doses (1 every 2.5 min)
- B. Four naloxone nasal spray doses (2 every 2.5 min) (Experimental): Four 4 mg IN naloxone doses (left and right nostrils at 0 min, left and right nostrils at 2.5 min)
  Interventions: Drug: Four naloxone nasal spray doses (2 every 2.5 min)
- C. Two naloxone nasal spray doses (1 every 2.5 min) (Active Comparator): Two 4 mg IN naloxone doses (left nostril at 0 min, right nostril at 2.5 min)
  Interventions: Drug: Two naloxone nasal spray doses (1 every 2.5 min)

INTERVENTIONS:
Drug: Four naloxone nasal spray doses (1 every 2.5 min) — Four 4 mg IN naloxone doses (left nostril at 0 min, right nostril at 2.5 min, left nostril at 5 min, right nostril at 7.5 min
  Other Names: Narcan nasal spray
  Arms: A. Four naloxone nasal spray doses (1 every 2.5 min)
Drug: Four naloxone nasal spray doses (2 every 2.5 min) — Four 4 mg IN naloxone doses (left and right nostrils at 0 min, left and right nostrils at 2.5 min)
  Other Names: Narcan nasal spray
  Arms: B. Four naloxone nasal spray doses (2 every 2.5 min)
Drug: Two naloxone nasal spray doses (1 every 2.5 min) — Two 4 mg IN naloxone doses (left nostril at 0 min, right nostril at 2.5 min)
  Other Names: Narcan nasal spray
  Arms: C. Two naloxone nasal spray doses (1 every 2.5 min)

SUMMARY:
Intranasal (IN) naloxone is available as 2 mg or 4 mg dose with the indication to re-administer additional doses every 2 to 3 minutes (using alternating nostrils) if needed until emergency medical assistance arrives. The 4 mg dose is distributed in packages of two nasal sprays (1 dose per nasal spray), but additional doses can be administered if needed and available.

While the pharmacokinetics of IN naloxone have been determined following administration of a 4 mg dose in each nostril concurrently, the pharmacokinetics have not been determined following multiple doses when there is a 2-3 minute delay between doses and when doses are re-administered to the same nostril.

Obtaining data with repeat dosing will inform if and how fast naloxone plasma concentrations can be reached to be able to reverse highly-potent opioid overdoses. This study will be a randomized, unblinded, three-way crossover study to determine naloxone plasma concentration after administration of multiple doses:

A. Four 4 mg IN naloxone doses (1 dose every 2.5 minutes) B. Four 4 mg IN naloxone doses (2 doses every 2.5 minutes) C. Two 4 mg IN naloxone doses (1 dose every 2.5 minutes)

DETAILED DESCRIPTION:
Naloxone, a fast-acting mu-opioid antagonist, is a treatment commonly used in reversing opioid overdose. Naloxone is available in multiple formulations, including for injection intravenously, intramuscularly or subcutaneously, and more recently as a spray administered intranasally (IN). The IN naloxone formulation, which was approved in 2015, is of particular interest as there is a need for naloxone formulations for community use by caregivers and first responders/law enforcement who do not have medical training. It is critical to administer naloxone as quickly as possible to prevent irreversible brain damage and death.

The U.S. Food and Drug Administration (FDA), Center for Drug Evaluation and Research (CDER), Division of Applied Regulatory Science (DARS) has conducted modeling and simulation, evaluating how many doses of IN naloxone may be needed to reverse opioid-induced respiratory depression from fentanyl and fentanyl derivates under a range of overdose scenarios. These analyses have suggested that more than two doses of IN naloxone are sometimes required to reverse the effects of highly potent opioids (e.g., certain fentanyl derivatives). Experience with intranasal formulations for other products has shown that repeat administration of doses given in close proximity to the same nostril can influence drug exposure due to run-off from the application site, limited absorption, or other factors. While the pharmacokinetics of IN naloxone have been determined following administration of a 4 mg dose in each nostril concurrently, the pharmacokinetics have not been determined following multiple doses according to the FDA product label:

* Administer a single spray intranasally into one nostril.
* Administer additional doses using a new nasal spray with each dose, if the patient does not respond or responds and then relapses into respiratory depression, additional doses may be given every 2 to 3 minutes until emergency medical assistance arrives.

This involves a 2-3 minute delay between each dose and re-administering to a previously dosed nostril starting with the 3rd dose, which may result in a less than dose-proportional increase in naloxone plasma concentration and/or delayed increase in naloxone exposure compared to the first 2 doses. Obtaining data with repeat dosing will inform if and how fast naloxone plasma concentrations can be reached to be able to reverse highly-potent opioid overdoses.

This study will be a randomized, unblinded, three-way crossover study to determine naloxone plasma concentration after administration of multiple doses:

A. Four 4 mg IN naloxone doses (1 dose every 2.5 minutes) B. Four 4 mg IN naloxone doses (2 doses every 2.5 minutes) C. Two 4 mg IN naloxone doses (1 dose every 2.5 minutes)

The above 3 treatments will be evaluated in a randomized order over 3 treatment periods. Healthy subjects will be randomized to one of six treatment sequences (i.e., ABC, ACB, BAC, BCA, CAB, CBA). Subjects will report to the study site for screening from Days -28 to -2 and then will return to the site on Day -1 for baseline assessments and check-in. After check-in (Day -1), subjects will receive dosing for the 3 respective treatment periods on Days 1, 4 and 7. There will be two days of washout between each treatment period. Participants will be confined in the study clinic from Day -1 until the morning of Day 8. On dosing days, dosing will occur as per the treatment description and pharmacokinetic (PK) assessments will occur at 16 different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an Institutional Review Board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization [HIPAA]) before any study related procedures are performed.
2. Subject is a healthy, non-smoking man or woman, 18 to 55 years of age, inclusive, who has a body mass index of 18.5 to 32 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead ECG results, and physical examination findings at screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and check-in (Day -1).
5. Subject must test negative for severe acute respiratory syndrome coronavirus (SARS-CoV-2) by a molecular diagnostic test at check-in (Day -1). If a subject's test comes back inconclusive, it can be repeated.
6. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before check-in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before check-in (Day -1) until at least 1 month after the end of the study.
7. Male subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee) from at least 1 month before check-in (Day -1) until at least 1 month after the last application of study drug.
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. Subject has a deviated septum or previous nasal surgeries or need to use another nasal spray product during study that would impact administration of the intranasal drug.
2. Subject has had an episode of epistaxis or an upper respiratory infection in the previous month.
3. Subject has used any prescription or nonprescription drugs (including aspirin or NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug.
4. Subject is currently participating in another clinical study of an investigational drug or has been dosed with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
5. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks of Screening.
6. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, cola), caffeine, grapefruit, or grapefruit juice within 24 h of check-in. Subjects must refrain from ingesting these throughout the study.
7. Subject has any underlying disease or surgical or medical condition (e.g., cancer, human immunodeficiency virus [HIV], severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study. This includes subjects with any underlying medical conditions that the Investigator believes would put subjects at increased risk of severe illness from COVID-19 based on the Centers for Disease Control and Prevention (CDC) guidelines. The CDC lists cancer, chronic kidney disease, chronic obstructive pulmonary disease, immunocompromised state from solid organ transplant, severe obesity, serious heart conditions, sickle cell disease, pregnancy, smoking and type 2 diabetes mellitus as conditions that put subjects at increased risk. Additionally, the CDC lists asthma (moderate-to-severe), cerebrovascular disease, cystic fibrosis, hypertension, immunocompromised state or immune deficiencies, neurologic conditions such as dementia, liver disease, pulmonary fibrosis, thalassemia, overweight, type 1 diabetes mellitus as conditions that might put subjects at increased risk.
8. Subject has any signs or symptoms that are consistent with COVID-19 per CDC recommendations. These include subjects with fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea may have COVID-19. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
9. Subject has known or suspected allergies or sensitivities to the study drug.
10. Subject has clinical laboratory test results (hematology, serum chemistry and urinalysis) at Screening or check-In that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
11. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
12. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or unlikely to complete the trial due to poor venous access.
13. Female subject is pregnant or lactating before enrollment in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Deering, MSN, APNP, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared at the time of the primary publication.
Supporting Information: Study Protocol, SAP
Time Frame: Individual patient data will be shared at the time of the primary publication, which is anticipated to be within 1 year of study completion.
Access Criteria: No restrictions.

REFERENCES:
- [Derived] Strauss DG, Li Z, Chaturbedi A, Chakravartula S, Samieegohar M, Mann J, Nallani SC, Prentice K, Shah A, Burkhart K, Boston J, Fu YA, Dahan A, Zineh I, Florian JA. Intranasal Naloxone Repeat Dosing Strategies and Fentanyl Overdose: A Simulation-Based Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2351839. doi: 10.1001/jamanetworkopen.2023.51839. PMID 38261323

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence ABC: Participants first received treatment A and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment A: Four 4 mg IN naloxone doses (1 dose every 2.5 min; Left nostril at 0 min, Right nostril at 2.5 min, Left nostril at 5 min, Right nostril at 7.5 min) Treatment B: Four 4 mg IN naloxone doses (2 doses every 2.5 min; Left and Right nostril at 0 min, Left and Right nostril at 2.5 min) Treatment C: Two 4 mg IN naloxone doses (Left nostril at 0 min, Right nostril at 2.5 min)
- Treatment Sequence ACB: Participants first received treatment A and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment A: Four 4 mg IN naloxone doses (1 dose every 2.5 min; Left nostril at 0 min, Right nostril at 2.5 min, Left nostril at 5 min, Right nostril at 7.5 min) Treatment C: Two 4 mg IN naloxone doses (Left nostril at 0 min, Right nostril at 2.5 min) Treatment B: Four 4 mg IN naloxone doses (2 doses every 2.5 min; Left and Right nostril at 0 min, Left and Right nostril at 2.5 min)
- Treatment Sequence BAC: Participants first received treatment B and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment B: Four 4 mg IN naloxone doses (2 doses every 2.5 min; Left and Right nostril at 0 min, Left and Right nostril at 2.5 min) Treatment A: Four 4 mg IN naloxone doses (1 dose every 2.5 min; Left nostril at 0 min, Right nostril at 2.5 min, Left nostril at 5 min, Right nostril at 7.5 min) Treatment C: Two 4 mg IN naloxone doses (Left nostril at 0 min, Right nostril at 2.5 min)
- Treatment Sequence BCA: Participants first received treatment B and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment B: Four 4 mg IN naloxone doses (2 doses every 2.5 min; Left and Right nostril at 0 min, Left and Right nostril at 2.5 min) Treatment C: Two 4 mg IN naloxone doses (Left nostril at 0 min, Right nostril at 2.5 min) Treatment A: Four 4 mg IN naloxone doses (1 dose every 2.5 min; Left nostril at 0 min, Right nostril at 2.5 min, Left nostril at 5 min, Right nostril at 7.5 min)
- Treatment Sequence CAB: Participants first received treatment C and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment C: Two 4 mg IN naloxone doses (Left nostril at 0 min, Right nostril at 2.5 min) Treatment A: Four 4 mg IN naloxone doses (1 dose every 2.5 min; Left nostril at 0 min, Right nostril at 2.5 min, Left nostril at 5 min, Right nostril at 7.5 min) Treatment B: Four 4 mg IN naloxone doses (2 doses every 2.5 min; Left and Right nostril at 0 min, Left and Right nostril at 2.5 min)
- Treatment Sequence CBA: Participants first received treatment C and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment C: Two 4 mg IN naloxone doses (Left nostril at 0 min, Right nostril at 2.5 min) Treatment B: Four 4 mg IN naloxone doses (2 doses every 2.5 min; Left and Right nostril at 0 min, Left and Right nostril at 2.5 min) Treatment A: Four 4 mg IN naloxone doses (1 dose every 2.5 min; Left nostril at 0 min, Right nostril at 2.5 min, Left nostril at 5 min, Right nostril at 7.5 min)
Period: Overall Study
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence CBA
Started | 3 | 4 | 3 | 4 | 3 | 4
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were randomized to 1 of 6 treatment sequences (i.e., ABC, ACB, BAC, BCA, CAB, CBA) and over 3 treatment periods received received 3 treatments as follows:
  Treatment A: Four 4 mg IN naloxone doses (1 dose every 2.5 min; Left nostril at 0 min, Right nostril at 2.5 min, Left nostril at 5 min, Right nostril at 7.5 min) Treatment B: Four 4 mg IN naloxone doses (2 doses every 2.5 min; Left and Right nostril at 0 min, Left and Right nostril at 2.5 min) Treatment C: Two 4 mg IN naloxone doses (Left nostril at 0 min, Right nostril at 2.5 min)
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 34 [27 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21
Body weight [Median (Inter-Quartile Range); unit: kg] | 79.6 [67.6 to 85.1]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.4 [24.8 to 30.6]

OUTCOME MEASURES:

1. Primary Outcome: First Timepoint When There is a Higher Naloxone Plasma Concentration in the 4 Naloxone Dose Arm (1 Every 2.5 Min) Compared to the 2 Naloxone Dose Arm (1 Every 2.5 Min)
Description: Naloxone plasma concentrations will be determined at specified timepoints. The four naloxone nasal spray dose arm (1 dose every 2.5 min) will be compared separately to the two naloxone nasal spray dose arm (1 dose every 2.5 min).
Time Frame: 10, 12.5, and 15 minutes, 10 minutes reported
Population: Includes any participant who had naloxone plasma concentration samples available within the specified PK sampling window and who did not miss one of the assigned doses. Prespecified timepoints for comparison were 10, 12.5, and 15 minutes. Only the data for the first timepoint when there is a higher naloxone plasma concentration in the 4 naloxone dose arm was prespecified for reporting. 10-minute data is shown. below
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 17 | 17
ng/mL | 8.49 (70) | 4.42 (159)
Statistical Analysis 1: Comparison: A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) vs C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min); Up to three different time points have been pre-specified for the comparison (10, 12.5, and 15 min). Time points will be evaluated from earliest to latest time. Testing will proceed until either one passes or all pre-specified time points fail. Subject-level naloxone concentrations will be log-transformed. Naloxone concentrations below the lower limit of quantification will result in that time point from that subject being removed for comparisons involving that treatment arm; Test type: Superiority — To demonstrate an increase in naloxone concentration, the lower bound of the one-sided 97.79% interval for the geometric mean ratio must exclude 1. The results will be transformed back to the original scale by exponentiation to provide treatment geometric means; p = 0.002, t-test, 1 sided — Testing will be conducted sequentially (i.e., start at the initial time and progress forward, stopping if success is achieved) at a 1-sided 0.0221 significance level since an increase in naloxone exposure is expected; Geometric mean ratio = 1.95, 95.6% CI 1-sided [lower limit 1.28] — Data is shown for 10-minute timepoint (first time point tested where an increased was observed). This compares results from the 4 naloxone dose arm (1 every 2.5 min) (numerator) with the 2 naloxone dose arm (1 every 2.5 min) (denominator); This was the first timepoint in the comparison that showed an increase in the 4 naloxone dose arm (1 every 2.5 min) compared to the 2 naloxone dose arm (1 every 2.5 min) and is the reported outcome for this endpoint

2. Primary Outcome: First Timepoint When There is a Higher Naloxone Plasma Concentration in the 4 Naloxone Dose Arm (2 Doses Every 2.5 Min) Compared to the 2 Naloxone Dose Arm (1 Every 2.5 Min)
Description: Naloxone plasma concentrations will be determined at specified timepoints. The four naloxone nasal spray dose arm (2 doses every 2.5 min) will be compared separately to the two naloxone nasal spray dose arm (1 dose every 2.5 min).
Time Frame: 4.5, 7, and 10 minutes
Population: Includes any participant who had naloxone plasma concentration samples available within the specified PK sampling window and who did not miss one of the assigned doses. Prespecified timepoints for comparison were 4.5, 7, and 10 minutes. Only the data for the first timepoint when there is a higher naloxone plasma concentration in the 4 naloxone dose arm (2 doses every 2.5 min) was prespecified for reporting. 4.5-minute data is shown. below
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 16 | 16
ng/mL | 2.24 (134) | 1.23 (250)
Statistical Analysis 1: Comparison: B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) vs C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min); Up to three different time points have been pre-specified for the comparison (4.5, 7, and 10 minutes). Time points will be evaluated from earliest to latest time. Testing will proceed until either one passes or all pre-specified time points fail. Subject-level naloxone concentrations will be log-transformed. Naloxone concentrations below the lower limit of quantification will result in that time point from that subject being removed for comparisons involving that treatment arm; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.018, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.98, 95.6% CI 1-sided [lower limit 1.03] — Data is shown for 4.5-minute timepoint (first time point tested where an increased was observed). This compares results from the 4 naloxone dose arm (2 doses every 2.5 min) (numerator) with the 2 naloxone dose arm (1 every 2.5 min) (denominator); This was the first timepoint in the comparison that showed an increase in the 4 naloxone dose arm (2 doses every 2.5 min) compared to the 2 naloxone dose arm (1 every 2.5 min) and is the reported outcome for this endpoint

3. Secondary Outcome: First Timepoint When There is a Higher Naloxone Plasma Concentration in the 4 Naloxone Dose Arm B (2 Doses Every 2.5 Min) Compared to the 4 Naloxone Dose Arm A (1 Dose Every 2.5 Minutes)
Description: Naloxone plasma concentrations will be determined at specified timepoints. The 4 naloxone dose arm B (2 doses every 2.5 min) will be compared to the 4 naloxone dose arm A (1 dose every 2.5 min)
Time Frame: 4.5, 7, and 10 minutes
Population: Includes any participant who had naloxone plasma concentration samples available within the specified PK sampling window and who did not miss one of the assigned doses. Prespecified timepoints for comparison were 4.5, 7, and 10 minutes. Only the data for the first timepoint when there is a higher naloxone plasma concentration in the 4 naloxone dose arm (2 every 2.5 min) was prespecified for reporting. 4.5-minute data is shown. below
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18
ng/mL | 2.24 (134) | 1.33 (124)
Statistical Analysis 1: Comparison: B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) vs A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min); [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.013, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.69, 95.6% CI 1-sided [lower limit 1.06] — Data is shown for 4.5-minute timepoint (first time point tested where an increased was observed). This compares results from the 4 naloxone dose arm (2 doses every 2.5 min) (numerator) with the 4 naloxone dose arm (1 every 2.5 min) (denominator); This was the first timepoint in the comparison that showed an increase in the 4 naloxone dose arm (2 doses every 2.5 min) compared to the 4 naloxone dose arm (1 every 2.5 min) and is the reported outcome for this endpoint

4. Secondary Outcome: Dose-proportionality of the 4 Naloxone Dose Arms in Reference to the 2 Naloxone Dose Arm Based on Maximum Concentration (Cmax).
Description: Dose proportionality based on Cmax will be compared between each of the three IN naloxone treatments as a secondary endpoint. For the comparisons, the 4 naloxone dose arms will be considered as the test and the reference will be the 2 naloxone dose arm. An additional comparison will be performed between the 4 naloxone dose arm B (2 doses every 2.5 min) as test and the 4 naloxone dose arm A (1 dose every 2.5 min) as reference. Values are reported as dose-normalized Cmax.
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, 30, 45, 60, 120, 180, 240, 360, and 720 minutes
Population: Includes any participant who receive study drug and have at least one post-dose sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL / mg (dose)
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL / mg (dose) | 1.10 (36) | 0.96 (44) | 1.25 (48)
Statistical Analysis 1: Comparison: A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) vs C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min); Dose-adjusted values for Cmax will be calculated based on noncompartmental PK parameter results, normalized to per mg of naloxone administered. Using linear mixed-effects modeling, comparisons of log-transformed dose-adjusted PK parameters will be performed. Treatment will be a fixed effect. Participant will be included as a random effect on the intercept; Test type: Other — Treatment differences on the log-scale will be estimated for the PK parameters. Geometric mean ratio and 90% CIs will be obtained by exponentiation of the treatment effect and 90% CIs based on the log-transformed scale. Dose-proportionality will be concluded if the confidence interval includes 1. Dose-normalized comparisons were exploratory; p = 0.10, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.89, 90% CI 2-sided [0.78 to 1.00] — This compares results from the 4 naloxone dose arm (1 every 2.5 min) (numerator) with the 2 naloxone dose arm (1 every 2.5 min) (denominator)
Statistical Analysis 2: Comparison: B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) vs C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min); [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.018, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.77, 90% CI 2-sided [0.65 to 0.92] — This compares results from the 4 naloxone dose arm (2 every 2.5 min) (numerator) with the 2 naloxone dose arm (1 every 2.5 min) (denominator)
Statistical Analysis 3: Comparison: A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) vs B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min); [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.12, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.87, 90% CI 2-sided [0.75 to 1.01] — This compares results from the 4 naloxone dose arm (2 every 2.5 min) (numerator) with the 4 naloxone dose arm (1 every 2.5 min) (denominator)

5. Secondary Outcome: Dose-proportionality of the 4 Naloxone Dose Arms in Reference to the 2 Naloxone Dose Arm Based on Area Under the Curve From Time 0 to Infinity (AUC0-inf)
Description: Dose proportionality based on AUC0-inf will be compared between each of the three IN naloxone treatments as a secondary endpoint. For the comparisons, the 4 naloxone dose arms will be considered as the test and the reference will be the 2 naloxone dose arm. An additional comparison will be performed between the 4 naloxone dose arm B (2 doses every 2.5 min) as test and the 4 naloxone dose arm A (1 dose every 2.5 min) as reference. Values are reported as dose-normalized AUC0-inf.
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, 30, 45, 60, 120, 180, 240, 360, and 720 minutes
Population: Includes any participant who received study drug and had at least one post-dose sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL * hr / mg (dose)
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL * hr / mg (dose) | 4.18 (25) | 3.79 (26) | 5.05 (21)
Statistical Analysis 1: Comparison: A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) vs B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min); Dose-adjusted values for AUC0-inf will be calculated based on noncompartmental PK parameter results, normalized to per mg of naloxone administered. Using linear mixed-effects modeling, comparisons of log-transformed dose-adjusted PK parameters will be performed. Treatment will be a fixed effect. Participant will be included as a random effect on the intercept; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.002, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.83, 90% CI 2-sided [0.76 to 0.91] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) vs C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min); [analysis description as in outcome 5, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p < 0.001, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.75, 90% CI 2-sided [0.70 to 0.81] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) vs B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min); [analysis description as in outcome 5, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.014, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.91, 90% CI 2-sided [0.85 to 0.97] — [estimate comment as in outcome 4, analysis 3]

6. Secondary Outcome: Dose-proportionality of the 4 Naloxone Dose Arms in Reference to the 2 Naloxone Dose Arm Based on Area Under the Curve From Time 0 to Last Sample (AUC0-t)
Description: Dose proportionality based on AUC0-t will be compared between each of the three IN naloxone treatments as a secondary endpoint. For the comparisons, the 4 naloxone dose arms will be considered as the test and the reference will be the 2 naloxone dose arm. An additional comparison will be performed between the 4 naloxone dose arm B (2 doses every 2.5 min) as test and the 4 naloxone dose arm A (1 dose every 2.5 min) as reference. Values are reported as dose-normalized AUC0-t.
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, 30, 45, 60, 120, 180, 240, 360, and 720 minutes
Population: Includes any participant who received study drug and had at least one post-dose sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL * hr / mg (dose)
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL * hr / mg (dose) | 4.13 (25) | 3.74 (26) | 5.05 (21)
Statistical Analysis 1: Comparison: A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) vs C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min); Dose-adjusted values for AUC0-t will be calculated based on noncompartmental PK parameter results, normalized to per mg of naloxone administered. Using linear mixed-effects modeling, comparisons of log-transformed dose-adjusted PK parameters will be performed. Treatment will be a fixed effect. Participant will be included as a random effect on the intercept; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.001, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.82, 90% CI 2-sided [0.75 to 0.89] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) vs C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min); [analysis description as in outcome 6, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p < 0.001, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.74, 90% CI 2-sided [0.69 to 0.80] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) vs B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min); [analysis description as in outcome 6, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.014, Mixed Models Analysis; Dose-normalized comparisons were exploratory; Geometric mean ratio = 0.91, 90% CI 2-sided [0.85 to 0.96] — [estimate comment as in outcome 4, analysis 3]

7. Secondary Outcome: Predicted Time to Rescue a Patient From Simulated Opioid-induced Respiratory Depression From Fentanyl for a Medium Overdose Scenario
Description: Data from this study will be combined with an existing pharmacokinetic/pharmacodynamic (PK/PD) model for opioid-induced respiratory depression to determine mean time to rescue. An intravenous fentanyl dose of 1.63 mg was selected as representative of a medium overdose scenario. The first naloxone dose in the simulations was administered 1 minute after ventilation decreased to 40% of baseline. Brain hypoxia (time to rescue a simulated patient) was defined as time brain oxygen partial pressure was less than 20 mm Hg and cardiac arrest was defined as the time cardiac output was less than 0.01 L/min. A value of 120 minutes means that simulated patients for that measure/dispersion metric were not predicted to recovered for the opioid dose and intervention.
Time Frame: 720 minutes
Population: Simulated patient data are reported as median and interquartile range (IQR) based on 200 randomly selected simulated patients from a population of 2000 with different pharmacokinetic and binding parameters and repeating this 2500 times with replacement. Reported result is the median and interquartile range from 2500 simulated studies with 200 simulated patients each.
Measure: Median (Inter-Quartile Range); unit: min
Units Other Than Participants: Number of Simulations
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 2000 | 2000 | 2000
Number analyzed (Number of Simulations) | 2500 | 2500 | 2500
min | 2.2 [0 to 4.5] | 1.6 [0 to 3.7] | 2.2 [0 to 4.5]

8. Secondary Outcome: Predicted Time to Rescue a Patient From Simulated Opioid-induced Respiratory Depression From Fentanyl for a High Overdose Scenario
Description: Data from this study will be combined with an existing pharmacokinetic/pharmacodynamic (PK/PD) model for opioid-induced respiratory depression to determine mean time to rescue. An intravenous fentanyl dose of 2.97 mg was selected as representative of a medium overdose scenario. The first naloxone dose in the simulations was administered 1 minute after ventilation decreased to 40% of baseline. Brain hypoxia (time to rescue a simulated patient) was defined as time brain oxygen partial pressure was less than 20 mm Hg and cardiac arrest was defined as the time cardiac output was less than 0.01 L/min. A value of 120 minutes means that simulated patients for that measure/dispersion metric were not predicted to recovered for the opioid dose and intervention.
Time Frame: 720 minutes
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: min
Units Other Than Participants: Number of Simulations
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 2000 | 2000 | 2000
Number analyzed (Number of Simulations) | 2500 | 2500 | 2500
min | 4.5 [2.1 to 120] | 3.7 [1.5 to 120] | 4.5 [2.1 to 120]

9. Secondary Outcome: Predicted Time to Rescue a Patient From Simulated Opioid-induced Respiratory Depression From Carfentanil for a Medium Overdose Scenario
Description: Data from this study will be combined with an existing pharmacokinetic/pharmacodynamic (PK/PD) model for opioid-induced respiratory depression to determine mean time to rescue. An intravenous carfentanil dose of 0.012 mg was selected as representative of a medium overdose scenario. The first naloxone dose in the simulations was administered 1 minute after ventilation decreased to 40% of baseline. Brain hypoxia (time to rescue a simulated patient) was defined as time brain oxygen partial pressure was less than 20 mm Hg and cardiac arrest was defined as the time cardiac output was less than 0.01 L/min. A value of 120 minutes means that simulated patients for that measure/dispersion metric were not predicted to recovered for the opioid dose and intervention.
Time Frame: 720 min
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: min
Units Other Than Participants: Number of Simulations
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 2000 | 2000 | 2000
Number analyzed (Number of Simulations) | 2500 | 2500 | 2500
min | 2.3 [0 to 120] | 1 [0 to 4.4] | 2.3 [0 to 120]

10. Secondary Outcome: Predicted Time to Rescue a Patient From Simulated Opioid-induced Respiratory Depression From Carfentanil for a High Overdose Scenario
Description: Data from this study will be combined with an existing pharmacokinetic/pharmacodynamic (PK/PD) model for opioid-induced respiratory depression to determine mean time to rescue. An intravenous carfentanil dose of 0.022 mg was selected as representative of a medium overdose scenario. The first naloxone dose in the simulations was administered 1 minute after ventilation decreased to 40% of baseline. Brain hypoxia (time to rescue a simulated patient) was defined as time brain oxygen partial pressure was less than 20 mm Hg and cardiac arrest was defined as the time cardiac output was less than 0.01 L/min. A value of 120 minutes means that simulated patients for that measure/dispersion metric were not predicted to recovered for the opioid dose and intervention.
Time Frame: 720 min
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: min
Units Other Than Participants: Number of Simulations
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 2000 | 2000 | 2000
Number analyzed (Number of Simulations) | 2500 | 2500 | 2500
min | 120 [4.1 to 120] | 120 [3.3 to 120] | 120 [4.1 to 120]

11. Other Pre Specified Outcome: Naloxone Cmax
Description: PK parameter for Cmax will be calculated
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, 30, 45, 60, 120, 180, 240, 360, and 720 minutes
Population: Includes any participant who received study drug and had at least one post-dose sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL | 17.6 (36) | 15.4 (44) | 10.0 (48)

12. Other Pre Specified Outcome: Naloxone AUC0-inf
Description: PK parameter AUC0-inf for naloxone will be calculated
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, 30, 45, 60, 120, 180, 240, 360, and 720 minutes
Population: Includes any participant who received study drug and had at least one post-dose sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL * hr
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL * hr | 1606 (25) | 1455 (26) | 978 (20)

13. Other Pre Specified Outcome: Naloxone AUC0-t
Description: PK parameter AUC0-t for naloxone will be calculated
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, 30, 45, 60, 120, 180, 240, 360, and 720 minutes
Population: Includes any participant who received study drug and had at least one post-dose sample collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL * hr
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL * hr | 1587 (25) | 1437 (26) | 970 (21)

14. Other Pre Specified Outcome: Naloxone Time of Maximum Concentration (Tmax)
Description: PK parameter tmax for naloxone will be calculated
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, 30, 45, 60, 120, 180, 240, 360, and 720 minutes
Population: Includes any participant who received study drug and had at least one post-dose sample collected.
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
min | 15 [15 to 20] | 15 [15 to 20] | 20 [15 to 30]

15. Other Pre Specified Outcome: Naloxone Partial Area Under the Curve (pAUC) From First Dose to 30 Minutes
Description: PK parameter pAUC from time 0 to 30 minutes for naloxone will be calculated
Time Frame: 0 [pre-dose], 2, 4.5, 7, 10, 12.5, 15, 20, and 30 minutes
Population: Includes any participant who received study drug and had at least one post-dose sample collected. Partial AUCs are reported for 0 minutes to 7 minutes, 0 minutes to 10 minutes, 0 minutes to 12.5 minutes, 0 minutes to 15 minutes, 0 minutes to 20 minutes, and 0 minutes to 30 minute.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL * hr
Arm/Group | A. Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | B. Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | C. Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL * hr
  Partial AUC 0 to 7.5 minutes | 9.2 (108) | 12.9 (121) | 6.0 (275)
  Partial AUC 0 to 10 minutes | 28.0 (87) | 34.6 (93) | 17.2 (176)
  Partial AUC 0 to 12.5 minutes | 54.1 (74) | 58.6 (87) | 28.8 (176)
  Partial AUC 0 to 15 minutes | 86.3 (68) | 93.9 (70) | 44.9 (137)
  Partial AUC 0 to 20 minutes | 162.7 (54) | 161.4 (57) | 84.0 (97)
  Partial AUC 0 to 30 minutes | 298.7 (40) | 279.5 (46) | 167.7 (37)

ADVERSE EVENTS:
Time Frame: 7 Days
Groups:
- Four Naloxone Nasal Spray Doses (1 Every 2.5 Min): Four 4 mg IN naloxone doses (left nostril at 0 min, right nostril at 2.5 min, left nostril at 5 min, right nostril at 7.5 min)
Arm/Group | Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) | Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) | Two Naloxone Nasal Spray Doses (1 Every 2.5 Min)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 11/21 | 5/21 | 8/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Four Naloxone Nasal Spray Doses (1 Every 2.5 Min) (N=21) | Four Naloxone Nasal Spray Doses (2 Every 2.5 Min) (N=21) | Two Naloxone Nasal Spray Doses (1 Every 2.5 Min) (N=21)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel Puncture Site Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Restless Leg Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (6) | 5 (8)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04764630/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT04764630/SAP_002.pdf
  • Informed Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT04764630/ICF_000.pdf